CLINICAL TRIAL: NCT00482833
Title: A Randomised Phase III Study to Compare Arsenic Trioxide (ATO) Combined to ATRA Versus Standard ATRA and Anthracycline-Based Chemotherapy (AIDA Regimen) for Newly Diagnosed, Non High-Risk Acute Promyelocytic Leukemia
Brief Title: Phase III Trial in Acute Promyelocytic Leukemia Patients
Acronym: APL0406
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Collaborators: Study Alliance Leukemia (SAL) Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL0406; GIMEMA-SAL-APL0406; EUDRACT-2006-006188-22
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Leukemia
Keywords: adult acute promyelocytic leukemia (M3); adult acute myeloid leukemia with t(15;17)(q22;q12); untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; Idarubicin; Mercaptopurine; Methotrexate; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A - ATO/ATRA (Experimental)
  Interventions: Drug: arsenic trioxide; Drug: all-trans retinoic acid (ATRA)
- ARM B - ATRA (Active Comparator)
  Interventions: Drug: idarubicin; Drug: mercaptopurine; Drug: methotrexate; Drug: all-trans retinoic acid

INTERVENTIONS:
Drug: arsenic trioxide — Induction Arsenic Trioxide (As2O3=ATO), 0.15 mg/Kg IV over 2 hours daily starting on day 1. ATO will be continued until hematological CR or for a maximum of 60 days.
  Consolidation ATO, 0.15 mg/Kg IV over 2 hours daily for 5 days every week. Treatment will be continued for 4 weeks on and 4 weeks off, for a total of 4 cycles (last cycle administered on weeks 25 - 28).
  Arms: ARM A - ATO/ATRA
Drug: idarubicin — Induction
  Idarubicin, 12 mg/m² on days 2, 4, 6 and 8 by short (20') intravenous infusion .
  If no hematological CR is achieved by 60 days after start of induction, patient will go off-study.
  Consolidation
  1st cycle Idarubicin, 5 mg/m2/day by short (20') intravenous infusion on days 1, 2, 3, 4.
  3rd cycle Idarubicin, 12 mg/m2/day as short (20') intravenous infusion only on day 1.
  Arms: ARM B - ATRA
Drug: mercaptopurine — Maintenance therapy 6-Mercaptopurine (6-MP), 50 mg/m2/day orally. The dose will be adjusted according to hematopoietic toxicity during the follow-up period
  Arms: ARM B - ATRA
Drug: methotrexate — Maintenance therapy Methotrexate (MTX), 15 mg/m2/weekly intramuscularly. The dose will be adjusted according to toxicity during the follow-up period.
  Arms: ARM B - ATRA
Drug: all-trans retinoic acid — Induction ATRA, 45 mg/m²/day will be administered orally in two equally divided doses and rounded to the nearest 10 mg increment, starting on day 1. ATRA treatment will be continued until hematological CR and for a maximum of 60 days.
  Consolidation
  1. st cycle ATRA, 45 mg/m2/day, will be administered orally in two equally divided doses and rounded to the nearest 10 mg increment, starting from day 1 to day 15.
  2. nd cycle ATRA, 45 mg/m2/day will be administered orally in two equally divided doses and rounded to the nearest 10 mg increment, starting from day 1 to day 15.
  3. rd cycle ATRA, 45 mg/m2/day will be administered orally in two equally divided doses and rounded to the nearest 10 mg increment, starting from day 1 to day 15.
  Maintenance therapy
  ATRA, 45 mg/m2/day orally, for 15 days every three months until a two year period is completed.
  Arms: ARM B - ATRA
Drug: all-trans retinoic acid (ATRA) — Induction All-trans retinoic acid (ATRA), 45 mg/m²/day will be administered orally in two equally divided doses and rounded to the nearest 10 mg increment, starting on day 1. ATRA treatment will be continued until hematological complete remission (CR, see below for definition) or for a maximum of 60 days.
  Consolidation ATRA, 45 mg/m²/day will be administered orally in two equally divided doses and rounded to the nearest 10 mg increment. Treatment will be administered for 2 weeks on 2 weeks off and for a total of 7 cycles (last cycle administered on weeks 25 - 26).
  Arms: ARM A - ATO/ATRA

SUMMARY:
Open label, randomised, phase III multicenter trial.

DETAILED DESCRIPTION:
* Arm I:

  * Induction therapy: Patients receive oral tretinoin twice daily and arsenic trioxide IV over 2 hours on days 1-60. Patients achieving hematological complete remission go on to receive consolidation therapy.
  * Consolidation therapy: Patients receive oral tretinoin twice daily on days 1-14. Treatment with tretinoin repeats every 4 weeks for up to 7 courses. Patients also receive arsenic trioxide IV over 2 hours on days 1-5 in weeks 1-4. Treatment with arsenic trioxide repeats every 8 weeks for up to 4 courses.
* Arm II:

  * Induction therapy: Patients receive tretinoin as in arm I induction therapy and idarubicin IV over 20 minutes on days 2, 4, 6, and 8. Patients achieving hematological complete remission go on to receive consolidation therapy.
  * Consolidation therapy: Patients receive oral tretinoin twice daily on days 1-45, idarubicin IV over 20 minutes on days 1-4 and day 31, and mitoxantrone hydrochloride IV over 30 minutes on days 16-20.

Marrow samples are collected after completion of consolidation therapy and analyzed by reverse transcriptase-PCR for molecular remission. Patients achieving molecular remission (PML-RARa negative) go on to receive maintenance therapy.

* Maintenance therapy: Patients receive oral mercaptopurine once daily and methotrexate intramuscularly once weekly for 3 months. Treatment with mercaptopurine and methotrexate repeats every 3 months for 7 courses. After completion of course 1 of mercaptopurine and methotrexate, patients receive oral tretinoin once daily on days 1-15*. Treatment with tretinoin repeats every 3 months for 6 courses.

NOTE: *Patients do not receive mercaptopurine and methotrexate during tretinoin administration.

After completion of study therapy, patients are followed periodically for 5 years.

As of 14th September 2010, all patients needed to evaluate the primary endpoint (162 patients) have been recruited but the trial accrual continued in order to assess one secondary outcome (QoL)."

ELIGIBILITY:
Inclusion criteria

* Signed written informed consent according to IGH/EU/GCP and national local laws
* Newly diagnosed APL by cytomorphology, confirmed also by molecular analysis*.
* Age ≤18 < 71 years
* WHO performance status 0 -2 included
* WBC at diagnosis ≤ 10 x 109/L
* Serum total bilirubin ≤ 3.0 mg/dL (≤ 51µmol/L)
* Serum creatinine ≤ 3.0 mg/dL (≤ 260 µmol/L)

The confirmation of diagnosis at genetic level (microspeckled PML nuclear distribution by PGM3 monoclonal antibody and/or PML/RARa fusion by RT-PCR and/or demonstration of t(15;17) by karyotyping) will be mandatory for patient eligibility. However, in order to avoid delay in treatment initiation, patients can be randomised on the basis of morphologic diagnosis only and before the results of genetic tests are available.

Exclusion criteria

* Age < 18 and ≥ 71
* WBC at diagnosis > 10 x 109/L
* Other active malignancy at time of study entry
* Lack of diagnostic confirmation at genetic level
* Significant arrhythmias, EKG abnormalities (*see below) or neuropathy
* Other cardiac contraindications for intensive chemotherapy (L-VEF <50%)
* Uncontrolled, life-threatening infections
* Severe non-controlled pulmonary or cardiac disease
* Women who are either pregnant or breast feeding, or of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they meet one of the following definitions:

  * Amenorrhea;
  * post surgical bilateral oophorectomy with or without hysterectomy;
  * using a highly effective method of birth control (defined as those which result in a failure rate less than 1% per year) when used consistently and correctly such as implants, injectables, oral contraceptives, IUDs, sexual abstinence or vasectomized partner.
* Concomitant severe psychiatric disorder
* HIV positivity

  *EKG abnormalities:
  * Congenital long QT syndrome;
  * History or presence of significant ventricular or atrial tachyarrhythmia
  * Clinically significant resting bradycardia (<50 beats per minute)
  * QTc > 450 msec on screening EKG (using the QTcF formula detailed on page 18)
  * Right bundle branch block plus left anterior hemiblock, bifascicular block
* Use of other investigational drugs at the time of enrolment or within 30 days before study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2007-08; Primary Completion 2012-09 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Event-free survival | At maximum 3.5 years from study entry
  As of 14th september 2010, all patients needed to evaluate the primary endpoint have been recruited.

SECONDARY OUTCOMES:
Rate of hematological complete remission | At maximum 60 days from induction therapy start
Overall survival rate | At 2 years from study entry
Rate of cumulative incidence of relapse | At 2 years from study entry
Incidence of hematological and non-hematological toxicity episodes during treatment as assessed by CTC-NCI | At maximum 60 days from induction therapy start and at maximum 225 days from consolidation therapy start
Rate of molecular remission after 3rd consolidation course | At maximum 225 days grom consolidation therapy start
Assessment of acute promyelocytic leukemia/RARa transcript level reduction after induction and during consolidation therapy | At maximum 60 days from induction therapy start and at maximum 225 days from consolidation therapy start
Quality of life at the end of induction therapy and at the end of the 3rd consolidation course | At maximum 60 days from induction therapy start and at maximum 225 days from consolidation therapy start
Event free survival | At 2 years from study entry
Total hospitalization days during study therapy | At maximum 3.5 years from study entry
Event-free survival rate in the two arms | At 2 years from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Lo Coco, MD, Study Chair — Azienda Ospedaliera Universitaria Policlinico Tor Vergata
Locations (110):
- Austria (3):
  - Universitätsklinik Innsbruck Hämatologie Onkologie, Innsbruck
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Universitätsklinik für Innere Medizin III Salzburg, Salzburg
- Germany (51):
  - Klinikum Bayreuth GmbH, Bayreuth
  - Charité Campus Benjamin Franklin Berlin, Berlin
  - Städt. Kliniken Bielefeld gem. GmbH, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Ev. Diakonie-Krankenhaus gGmbH Bremen, Bremen
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum C. G. Carus Dresden, Dresden
  - Katholisches Klinikum Duisburg St. Johannes Hospital, Duisburg
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Uniklinikum Erlangen, Erlangen
  - Kliniken Essen Süd, Ev. Krankenhaus Essen-Werden gGmbH, Essen
  - Universitätsklinikum Essen, Essen
  - Uniklinik Frankfurt/Main, Frankfurt am Main
  - Städtische Kliniken Frankfurt a. M.-Höchst, Frankfurt/a. M. -Höchst
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Fulda, Fulda
  - Universitätsklinikum Gießen und Marburg Gießen, Giessen
  - Universitätsklinikum Göttingen, Göttingen
  - Asklepios Klinik Hamburg Altona, Hamburg
  - Asklepios Klinik St. Georg Hamburg, Hamburg
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - St. Marien-Hospital gem. GmbH Hamm, Hamm
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - St. Bernward Krankenhaus Hildesheim, Hildesheim
  - Universitätsklinikum des Saarlandes Homburg/Saar, Homburg
  - Klinik für Knochenmarktransplantation und Hämatologie Idar-Oberstein, Idar-Oberstein
  - Westpfalz-Klinikum GmbH Kaiserslautern, Kaiserslautern
  - Caritas-Krankenhaus Lebach, Lebach
  - Klinikum Lippe Lemgo, Lippe
  - Uniklinikum Lübeck, Lübeck
  - Klinikum der Johannes Gutenberg Universität Mainz, Mainz
  - Universitätsklinikum Gießen und Marburg GmbH Marburg, Marburg
  - Carl-von-Basedow-Klinikum Merseburg, Merseburg
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum rechts der Isar (München), München
  - Klinikum Nord Nürnberg, Nuremberg
  - Klinikum Passau, Passau
  - Universitätsklinikum Regensburg, Regensburg
  - Caritas-Klinik St. Theresia Saarbrücken, Saarbrücken
  - Diakonie-Krankenhaus Schwäbisch Hall, Schwäbisch Hall
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Klinikum Stuttgart Bürgerhospital, Stuttgart
  - Robert Bosch Krankenhaus Stuttgart, Stuttgart
  - Krankenanstalt Mutterhaus der Borromäerinnen Trier, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Villingen-Schwenningen, Villingen-Schwenningen
  - HELIOS Klinikum Wuppertal, Wuppertal
- Italy (56):
  - Ospedale Civile SS. Antonio e Biagio di Alessandria, Alessandria
  - Ospedale Gen.le. Prov.le "C.G. Mazzoni", Ascoli Piceno
  - Az.Ospedaliera S.G.Moscati, Avellino
  - Ematologia con trapianto- AOU Policlinico Consorziale di Bari, Bari
  - Divisione di Ematologia - Ospedali Riuniti, Bergamo
  - Istituto di Ematologia e Oncologia Medica "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Sanitaria di Bolzano - Ospedale Centrale - Ematologia e Centro TMO, Bolzano
  - Spedali Civili di Brescia, Brescia
  - ASL N.8 - Ospedale "A. Businco" - Unità Operativa di Ematologia e Trapianto di Midollo, Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Sezione di Ematologia e Fisiopatologia delle Emostasi - Azienda Ospedaliera - Arcispedale S. Anna, Ferrara
  - Divisione Ematologia 1 - Azienda Ospedaliera Universitaria "San Martino", Genova
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - ST. V. Fazzi, Lecce
  - A.O. Universitaria Policlinico Martina di Messina, Messina
  - Azienda ospedaliera Papardo, Messina
  - IRCCS Fondazione Centro S. Raffaele del Monte Tabor, Milan
  - Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Milan
  - UO Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - Azienda ospedaliera S. Gerardo di Monza, Monza
  - A.S.L. Napoli 1 Ospedale San Giovanni Bosco, Napoli
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Servizio Sanitario Nazionale - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli" - Struttura Complessa di Ematologia - Div. TERE- 4° piano - Padiglione Palermo, Napoli
  - ASL SA/1 di Nocera Inferiore, Nocera Inferiore
  - A.O. Universitaria S. Luigi Gonzaga di Orbassano, Orbassano
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - IRCCS Policlinico S. Matteo di Pavia, Pavia
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della MIsericordia, Perugia
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Ematologia - Ospedale San Carlo, Potenza
  - Ospedale S. Maria delle Croci di Ravenna, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - IRCCS Centro di riferimento Oncologico di Basilicata, Rionero in Vulture
  - Azienda Osp. S. Giovanni/Addolorata, Roma
  - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - Ospedale S. Eugenio, Roma
  - Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Policlinico Campus Biomedico, Roma
  - Policlinico Universitario Gemelli di Roma, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - IRCCS Istituto Regina Elena, Rome
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Serv. di Ematologia Ist. di Ematologia ed Endocrinologia, Sassari
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - SCDO Ematologia 2 AOU S.Giovanni Battista, Torino
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Ospedale di circolo e Fondazione Macchi, Varese
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona
  - ULSS N.6 Osp. S. Bortolo, Vicenza

REFERENCES:
- [Derived] Efficace F, Mandelli F, Avvisati G, Cottone F, Ferrara F, Di Bona E, Specchia G, Breccia M, Levis A, Sica S, Finizio O, Kropp MG, Fioritoni G, Cerqui E, Vignetti M, Amadori S, Schlenk RF, Platzbecker U, Lo-Coco F. Randomized phase III trial of retinoic acid and arsenic trioxide versus retinoic acid and chemotherapy in patients with acute promyelocytic leukemia: health-related quality-of-life outcomes. J Clin Oncol. 2014 Oct 20;32(30):3406-12. doi: 10.1200/JCO.2014.55.3453. Epub 2014 Sep 22. PMID 25245446
- [Derived] Lo-Coco F, Avvisati G, Vignetti M, Thiede C, Orlando SM, Iacobelli S, Ferrara F, Fazi P, Cicconi L, Di Bona E, Specchia G, Sica S, Divona M, Levis A, Fiedler W, Cerqui E, Breccia M, Fioritoni G, Salih HR, Cazzola M, Melillo L, Carella AM, Brandts CH, Morra E, von Lilienfeld-Toal M, Hertenstein B, Wattad M, Lubbert M, Hanel M, Schmitz N, Link H, Kropp MG, Rambaldi A, La Nasa G, Luppi M, Ciceri F, Finizio O, Venditti A, Fabbiano F, Dohner K, Sauer M, Ganser A, Amadori S, Mandelli F, Dohner H, Ehninger G, Schlenk RF, Platzbecker U; Gruppo Italiano Malattie Ematologiche dell'Adulto; German-Austrian Acute Myeloid Leukemia Study Group; Study Alliance Leukemia. Retinoic acid and arsenic trioxide for acute promyelocytic leukemia. N Engl J Med. 2013 Jul 11;369(2):111-21. doi: 10.1056/NEJMoa1300874. PMID 23841729
- See also: GIMEMA Foundation Website — http://www.gimema.it